CLINICAL TRIAL: NCT04076930
Title: Effects of Renin-Angiotensin System Inhibitors on Mortality and Cardiovascular Outcomes in Peritoneal Dialysis Patients: A Retrospective Cohort Study in Thailand
Brief Title: Effects of Renin-Angiotensin System Inhibitors in Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Chidchanok Ruengorn, Principal Investigator, Chiang Mai University
Other Study IDs: THOR-PD: RAS Inhibitors
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Peritoneal Dialysis
Keywords: Cardiovascular; Hyperkalemia; Mortality; Peritoneal dialysis; Renin-angiotensin system; Retrospective cohort
MeSH Terms: conditions — Hyperkalemia | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ACEI/ARB users
  Interventions: Drug: angiotensin-converting enzyme inhibitor (ACEI) and angiotensin receptor blocker (ARB)
- ACEI/ARB non-users

INTERVENTIONS:
Drug: angiotensin-converting enzyme inhibitor (ACEI) and angiotensin receptor blocker (ARB) — The use of ACEI/ARB within a 90-day after the date of PD initiation (exposure ascertainment window period).
  Groups: ACEI/ARB users

SUMMARY:
Among antihypertensive medications, RAS inhibitor classes, namely angiotensin-converting enzyme inhibitor (ACEI) and angiotensin receptor blocker (ARB) have the most prospective data on mortality and cardiovascular outcomes in specific high-risk populations with mild to moderate chronic kidney disease (CKD). Whereas, long-term data on the risks and benefits of ACEI/ARB usage in end-stage kidney disease (ESKD) patients undergoing peritoneal dialysis (PD) are limited. Recently, increasing clinical studies suggested that ACEI/ARB had a beneficial effect on intermediate outcomes, including short-term blood pressure variability, left ventricular hypertrophy, and may have an important role in the peritoneum and the kidney protection. Subsequently, treatment with ACEI/ARB has been recommended by the International Society for Peritoneal Dialysis for PD patients with significant residual kidney function (RKF).

Although existing reviews demonstrated that ACEI/ARB significantly has benefit in preserving RKF in PD patients, evidence regarding the relative efficacy on mortality, cardiovascular outcomes, and adverse events is lacking. Given that there exist few controlled trials of the effectiveness of ACEI/ARB in PD patients, we intend to perform a retrospective cohort study to assess the association between the use of ACEI/ARB and the risk of long-term mortality, cardiovascular outcomes, and adverse events in terms of hyperkalemia.

A retrospective cohort of Thai PD patients will be constructed by using the local joint registry data of adult PD patients from five centers in Thailand between 2006 to 2017 and followed to December 2018. We will link the following health datasets: (i) the electronic health records, contains outpatient and inpatient data; (ii) the Support System Pharmacy Dispensing extract, an administrative database which covers pharmacy dispensing; (iii) the PD Patient Care Database, which provides patient-level detail on sociodemographic and clinical characteristics as well as long-term PD care data; and (iv) the Laboratory Support System extract, which includes claims and routine laboratory results.

The exposure of interest in this cohort will be the use of ACEI/ARB within a 90-day after the date of PD initiation. Outcomes of interest will include all-cause mortality, cardiovascular mortality, a composite endpoint of cardiovascular events, and adverse events in terms of hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or over at the date of PD initiation
* Patients with ESKD who were undergoing PD either continuous ambulatory peritoneal dialysis or automated peritoneal dialysis between January 1, 2006, to December 31, 2017
* Received PD treatment more than 90 days in an outpatient nephrology clinic visit after the date of PD initiation
* Received of any outpatient prescriptions within 90 days after the date of PD initiation

Exclusion Criteria:

* Previously been treated by maintenance hemodialysis (for more than 90 days) or initiated PD for acute kidney injury or after a failed kidney transplantation
* Died within 90 days after the date of PD initiation
* Received a combination of ACEIs and ARBs therapy
* Received ACEIs/ARBs within 180 days before PD initiation
* Had no information regarding ACEI/ARB dosage regimen during the follow-up period
* Inadequate follow-up clinical information on blood pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ESKD patients undergoing PD from January 1, 2006, to December 31, 2017, and followed to December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1468 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 years
Cardiovascular mortality | 12 years

SECONDARY OUTCOMES:
Composite endpoint of atherosclerotic cardiovascular disease (ASCVD) events | 12 years
  ASCVD events of interest will include hospitalization for acute fatal and nonfatal myocardial infarction, coronary or other arterial revascularization, fatal and nonfatal stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin.
Hyperkalemia | 12 years
  Incident hyperkalemia will define as a serum potassium concentration of more than 5.0 mEq/L. The severity of hyperkalemia will be categorized as mild (>5.0 to <5.5 mEq/L), moderate (5.5 to 6.0 mEq/L), and severe (>6.0 mEq/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacoepidemiology and Statistics Research Center, Faculty of Pharmacy, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data from the retrospective cohort study part will be made available at the end of the study, on request. Requests will subject to approval by the chief investigator, the advisory Committee and the relevant ethical bodies.